CLINICAL TRIAL: NCT04742725
Title: A Randomized, Double Blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Prothione™ Capsules for Mild to Moderate Coronavirus Disease 2019 (COVID-19)
Brief Title: A Study to Evaluate the Efficacy and Safety of Prothione™ Capsules for Mild to Moderate Coronavirus Disease 2019 (COVID-19)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prothione, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAL-PRO-001
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Coronavirus Disease 2019 (COVID-19)
Keywords: COVID-19, Prothione
MeSH Terms: conditions — COVID-19 | interventions — Prothione

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Prothione ™ (Experimental)
  Interventions: Drug: Prothione™ (6g)

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Prothione™ (6g) — Prothione is a pro-Glutathione compound includes free-form amino acids
  Arms: Prothione ™

SUMMARY:
The study is a phase 2 proof of concept study. The purpose of this study is to assess the efficacy and safety of Prothione™ capsules administered orally twice a day for 30 days in subjects with mild to moderate COVID-19. The study will have three phases: Screening Period, Treatment Period, and Follow-Up Period.

The issued patents relevant to Prothione™ capsules and the treatment of viral disease include: • Nutritional or Therapeutic Compositions and Methods to Increase Bodily

Glutathione Levels:

1. US Patent No. RE 42,645
2. Japanese Patent No. 5601745
3. European Patent No. 1556023
4. Canadian Patent No. 2539567
5. Australian Patent No. 2010201136

   • Protective Metallothionein Analog Compounds, Their Compositions and Use

   Thereof in the Treatment of Pathogenic Disease:
6. Canadian Patent No. 2963131
7. Australian Patent No. 2018279015

DETAILED DESCRIPTION:
This is a Phase 2, proof of concept, two-arm, randomized, double blind, placebo-controlled study to evaluate the safety and efficacy of Prothione™ capsules in subjects with mild-to-moderate symptoms caused by coronavirus 2019 (COVID-19) infection. Subjects will be randomized to receive three Prothione™ capsules, or placebo orally administered twice daily (BID).

The study will have three phases: screening period, treatment period, and follow-up period. Screening period is up to 3 days , the treatment period is 30 days and the follow-up period is 7 days after the last dose.Total study duration is up to 40 days.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects are required to meet all of the following criteria for enrollment into the study:

1. Male or female adult ≥ 18 years of age at time of enrollment with mild to moderate symptoms caused by coronavirus 2019 confirmed infection with COVID-19 by PCR and one or more of the following:

   Mild (uncomplicated) Illness:
   * Diagnosed with COVID-19 by a standardized RT-PCR assay AND
   * Mild symptoms, such as fever, rhinorrhea, mild cough, sore throat, malaise, headache, muscle pain, or malaise, but with no shortness of breath AND
   * No signs of a more serious lower airway disease AND RR<20, HR <90, oxygen saturation (pulse oximetry) > 93% on room air

   Moderate Illness:
   * Diagnosed with COVID-19 by a standardized RT-PCR assay AND
   * In addition to symptoms above, more significant lower respiratory symptoms, including shortness of breath (at rest or with exertion) OR
   * Signs of moderate pneumonia, including RR ≥ 20 but <30, HR ≥ 90 but less than 125, oxygen saturation (pulse oximetry) > 93% on room air AND
   * If available, lung infiltrates based on X-ray or CT scan < 50% present
2. Subjects with normal level of Vitamin B2; Note: If the result was below the normal range, based on clinical judgment by physician, appropriate treatment to be added to the subject treatment regimen as per standard of care. A B complex daily supplement will be supplied, if needed.
3. Subject (or legally authorized representative) provides written informed consent prior to initiation of any study procedures;
4. Understands and agrees to comply with planned study procedures; and
5. Negative pregnancy test for female subjects. Women of child-bearing potential (WOCBP) and Women not of child-bearing potential are eligible to participate. Both women of child-bearing potential and women of no child-bearing potential should use an approved method of birth control and agrees to continue to use this method for the duration of the study (and for 30 days after taking the last dose of Prothione™ ).

Acceptable methods of contraception include abstinence, female subject/partner's use of hormonal contraceptive (oral, implanted, or injected) in conjunction with a barrier method (WOCBP only), female subject/partner's use of an intrauterine device (IUD), or if the female subject/partner is surgically sterile or 2 years post-menopausal. All male subjects/partners must agree to consistently and correctly use a condom for the duration of the study. In addition, subjects may not donate sperm for the duration of the study and for 30 days after taking study drug.

Exclusion Criteria:

Potential subjects meeting any of the following criteria will be excluded from enrollment:

1. Subjects showing signs of acute respiratory distress syndrome (ARDS) or respiratory failure necessitating mechanical ventilation at the time of screening;
2. Subjects who have history of receiving NAC, Prothione™ Capsules or GSH supplements in the past 30 days before the screening visit;
3. Subjects who have history of receiving corticosteroids (topical corticosteroid is excluded) in the past 30 days;
4. Subjects who are currently receiving Chemotherapy or Immunotherapy for the treatment of cancer;
5. Any uncontrolled active systemic infection requiring admission to an intensive care unit (ICU);
6. Subject with active Hepatitis B and Hepatitis C;
7. Subjects who are participating in other clinical trials;
8. Subjects that have had any Covid19 Vaccination;
9. Subjects who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to Prothione™ are not eligible;
10. Inability to provide informed consent or to comply with study requirements; and
11. Subjects who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Time (days) to successful clinical recovery from positive RT-PCR for SARS-COV2 as indicated by two consecutive negative RT-PCR tests measured with three different measurements within a 24-36 hour period. | 24-36 hour period

SECONDARY OUTCOMES:
Change from Baseline to Day 29 in Serum 8-OHdG levels | Baseline to day 29
Change in RBC intracellular Glutathione levels to Day 29 | Baseline to day 29
Quantitative change from Baseline (Screening Visit) to Day 29 oropharyngeal cell intracellular GSH levels | Baseline to day 29
Time to clinical resolution (TTCR) defined as the time (days) from initiation of study treatment until reach a score of 0 at least in three of the following: o Fever o Myalgia o Dyspnea o Cough | Baseline to day 29
  ( Each symptom is graded from 0 to 3. [0=none 1=mild 2=moderate and 3=severe]
Evaluate Cycle Threshold (Ct) numbers used in qualitative and quantitative RT-PCR for SARS-COV2 tests. | Baseline to day 29
Clinical Improvement as assessed by change in symptom score from baseline (for fever, myalgia, dyspnea and cough). | Baseline to day 29
  Note: The score per patient ranges from 0 to 3 points. Each symptom is graded from 0 to 3. [0=none, 1=mild, 2=moderate, and 3=severe]
Mortality at Day 29 | Day 29

OTHER OUTCOMES:
Quantitative changes in viral load from baseline (Screening Visit) to Day 29. | Baseline to day 29
  Exploratory Outcome
Change from baseline to Day 29 in pulse oxygen saturation (SpO2) | Baseline to day 29
  Exploratory Outcome
Change from baseline to Day 29 in Quantitative C-Reactive Protein level | Baseline to Day 29
  Exploratory Outcome
Change from baseline to Day 29 in Lymphocyte Count | Baseline to Day 29
  Exploratory Outcome
Changes in HIV viral load from baseline to Day 29 in HIV positive subjects | Baseline to Day 29
  Exploratory Outcome
Duration (days) of hospitalization | Baseline to Day 29
  Exploratory Outcome
Time(days) to clinical resolution (TTCR) before Day 14 | Before Day 14
  Exploratory Outcome
Time (days) to successful clinical recovery from positive RT-PCR for SARS-COV2 as indicated by three consecutive negative RT-PCR tests measured with two different measurements within a 24-36 hour period before Day 14. | within a 24-36 hour period before Day 14
  Exploratory Outcome
Quantitative changes in viral load from baseline (Screening Visit) to Day 14 | Baseline to Day 14
  Exploratory Outcome
Change from baseline to Day 14 in Quantitative C-Reactive Protein level | Baseline to Day 14
  Exploratory Outcome
Incidence of treatment-related adverse events (TEAEs) | until day 40
  Safety Outcome
Incidence and severity of treatment-emergent adverse events (TEAEs) | until day 40
  Safety Outcome
Incidence of serious adverse events (SAEs) | until day 40
  Safety Outcome
Incidence of TEAEs and SAEs leading to discontinuation of study medication. | until day 40
  Safety Outcome
Incidence of abnormal laboratory test results | until day 40
  Safety Outcome
Changes in body temperature | until day 40
  Safety Outcome
Changes in pulse rate | until day 40
  Safety Outcome
Changes in respiratory rate | until day 40
  Safety Outcome
Changes in systolic and diastolic blood pressure | until day 40
  Safety Outcome
Incidence of abnormal physical examination findings | until day 40
  Safety Outcome
Incidence of abnormal electrocardiogram (ECG) results | until day 40
  Safety Outcome

CONTACTS AND LOCATIONS:
Overall Officials: Laura Lile, MD,RPh, Principal Investigator — Innate FFAAP Medicines, L.L.C.; Vincent Mutabazi, MD, Principal Investigator — Research, Epidemiology and Training Programs: RASD Rwanda; Albert Crum, MD, Study Chair — Innate FFAAP Medicines, L.L.C.
Locations (1):
- Rinda Ubuzima, Kigali, Rwanda